CLINICAL TRIAL: NCT07185048
Title: Clinical AI-powered Remote Engagement for Diabetic Foot Ulcer Prevention
Brief Title: Evaluation of the Clinical Efficacy and Feasibility of Digital Foot Care Intervention Strategies With Different Intensities in the Prevention of Diabetic Foot Ulcers.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-302
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcers (DFUs)
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Foot Care Control Group (Active Comparator)
  Interventions: Behavioral: Conventional Foot Care Control Group
- Low-Intensity Digital Foot Care Group (Experimental)
  Interventions: Behavioral: Digital Foot Care (Low-Intensity)
- Moderate-Intensity Digital Foot Care Group (Experimental)
  Interventions: Behavioral: Digital Foot Care (Moderate-Intensity)

INTERVENTIONS:
Behavioral: Conventional Foot Care Control Group — Standard Foot Care with Regular Follow-up
  Arms: Conventional Foot Care Control Group
Behavioral: Digital Foot Care (Low-Intensity) — On the basis of routine management, the digital intervention modules will be added
  Arms: Low-Intensity Digital Foot Care Group
Behavioral: Digital Foot Care (Moderate-Intensity) — Further integration of AI image analysis for auxiliary judgment and remote physician response.
  Arms: Moderate-Intensity Digital Foot Care Group

SUMMARY:
For people with diabetes who are at risk of foot ulcers, this study compares three digital foot care strategies (with different levels of intensity) to see which one is more effective at preventing ulcers and easier to use.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years but < 80 years;
2. Assessed to meet the criteria for the high-risk population for diabetic foot as defined by the International Working Group on the Diabetic Foot (IWGDF) (risk level 3);
3. Capable of using a smartphone to take photos and operate apps, or able to do so after simple training;
4. Willing to participate in the study and sign an informed consent form.

Exclusion Criteria:

1. Currently has an open foot wound or an unresolved foot ulcer;
2. History of major lower limb amputation above the ankle joint;
3. Pregnancy or breastfeeding;
4. Currently suffering from poorly controlled malignant tumors;
5. Receiving glucocorticoid or immunosuppressive therapy;
6. Diagnosed with vascular occlusive vasculitis;
7. Presence of foot fracture;
8. Significant visual impairment affecting image acquisition or operation;
9. Other conditions deemed inappropriate for participation in this study by the research team.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1512 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Diabetic Foot Ulcers | 18 months after intervention initiation

IPD SHARING:
Plan to Share IPD: No